CLINICAL TRIAL: NCT06128694
Title: The Effect of Oral Nutrition Supplement Formulas (ONS) and Diet Counseling on Improvement of Nutritional Status, Knowledge, Attitudes, and Behavior of Cancer Patients
Brief Title: Effect of NUTRICAN to Improve Nutritional Status in Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kalbe International Pte. Ltd (Industry)
Collaborators: Persahabatan Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Constatine Study
Record Dates: First submitted 2023-10-23; First posted 2023-11-13 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-11

CONDITIONS: Malnutrition; Protein; Cancer, Lung; Cancer Cervix
Keywords: malnutrition; oral nutrition supplement; cancer; Nutrican
MeSH Terms: conditions — Kwashiorkor; Lung Neoplasms; Uterine Cervical Neoplasms; Malnutrition; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONS (oral nutrition supplement) group (Experimental): ONS will be consumed 3 times a day, for 8 weeks. Per serving/sachet ONS (±81g) contains 350 kcal of energy, 9 g of fat, 20 g of protein, 48 g of carbohydrates, 400 mg of DHA (Docosahexaenoic acid), 300 mg of EPA (Eicosapentaenoic Acid) 0.92 g of Omega-3, 1 g of L-Valine, 2.1 g of L-. Isoleucine 1.1 g, L-Leucine 2.1 g, Sodium 75 mg, 12 vitamins and 9 minerals. Consumed as a morning snack (between breakfast and lunch); afternoon snack (between lunch and dinner) and evening snack (before bedtime). Subject will also received dietary counseling for 8 weeks
  Interventions: Dietary Supplement: NUTRICAN
- Control group (No Intervention): only received dietary counseling for 8 weeks without ONS supplementation.

INTERVENTIONS:
Dietary Supplement: NUTRICAN — Per serving/sachet NUTRICAN (±81g) contains 350 kcal energy, 9 g fat, 20 g protein, 48 g carbohydrate, 400 mg DHA, 300 mg EPA, 0.92 g Omega-3, 1 g L-Valine, 1.1 g L-Isoleucine, 2.1 g L-Leucine, 75 mg sodium, 12 vitamins and 9 minerals.
  Arms: ONS (oral nutrition supplement) group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy oral nutrition supplement (ONS) in malnutrition/high risk malnutrition cancer patients. The main questions it aims to answer:

1. Are there differences in knowledge, attitude and behaviour scores in cancer patients who receive cancer-specific ONS compared to those who do not receive cancer-specific ONS?
2. Is there a difference in nutritional status as assessed by average body weight, body mass index (BMI), haemoglobin (Hb), and albumin levels in cancer patients who receive cancer-specific ONS compared to those who do not receive cancer-specific ONS?

DETAILED DESCRIPTION:
This study uses an open label randomized clinical trial (RCT) design, double arm which allows subjects and researchers to know the interventions received by subjects conducted on cancer patient subjects. The study aims to compare knowledge, attitudes, and actions related to nutrition consumption through questionnaires, nutritional status assessed from anthropometry (BW and BMI), nutrient intake, as well as laboratory results (Hb, serum albumin), and inflammatory markers (CRP, TNF-α, IL(interleukin)-1, IL-6) between the group of subjects who were given dietary counseling and ONS/oral nutrition supplement (intervention group) for 8 weeks compared to the group of subjects who only received dietary counseling and did not receive ONS (control group).

Subjects who meet the inclusion criteria will be randomized into 2 groups using the stratified block randomization method stratified by age, and cancer type. Randomization will be carried out using a system in the application by stratifying the age of the subject based on the categorical age which has been categorized into 18-45 years and >45 years. For the type of cancer stratified into two, namely lung cancer and gynecology cancer according to the inclusion criteria. Both stratified will be randomized using excel application that will randomize 80 subjects at the beginning of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed lung and ob-gyn cancer patients (who have not undergone therapy or are currently undergoing therapy)
* Aged greater than or equal to 18 years
* Patients with a performance status score of 0 - 2
* Have inadequate food intake >5 days or:

  1. BMI/body mass index <18.5 kg/m2 or
  2. There is a >10% weight loss in the last 3-6 months or
  3. BMI <20 kg/m2 or
  4. There is >5% weight loss in the last 3-6 months with
* Intervention group subjects are willing to take ONS orally for 8 weeks
* Intervention group subjects, if they have taken other brands of ONS, are willing to stop taking ONS 2 weeks prior to the study.

Exclusion Criteria:

* Pregnant and breastfeeding, except for female subjects with one of the following criteria:

  1. Have a history of hysterectomy (surgical removal of the uterus) and/or bilateral oophorectomy (surgical removal of the ovaries).
  2. Medically confirmed ovarian failure (decreased ovarian function)
  3. Achieved post menopausal status, defined as: cessation of regular menstruation for at least 12 consecutive months in the absence of pathological or physiological causes.
* Renal insufficiency (eGFR ( Estimated Glomerular Filtration Rate ) <15 mL/min/1.73 m2 or significant increase in urea/creatinine or having to be on a low protein diet)
* Liver insufficiency (SGOT (Serum Glutamic Oxaloacetic Transaminase) /SGPT (Serum Glutamic Pyruvic Transaminase) values ≥3 times the normal limit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Nutrition consumption knowledge score | 8 weeks
  To determine changes in nutrition consumption knowledge scores in cancer patients who received cancer-specific ONS compared to those who did not receive ONS after 8 weeks of intervention using questioner .
  Interpretation Knowledge score (5 questions): good (score>=8 ) moderate (score 5-8) poor (score 0-4);
Nutrition consumption attitude score | 8 weeks
  To determine changes in nutrition consumption attitudes score in cancer patients who received cancer-specific ONS compared to those who did not receive ONS after 8 weeks of intervention using questioner .
  Interpretation Attitude score (10 questions): good (score>=30 ) moderate (score 21-30) poor (score 0-20)
Nutrition consumption behaviour score | 8 weeks
  To determine changes in nutrition consumption behavior in cancer patients who received cancer-specific ONS compared to those who did not receive ONS after 8 weeks of intervention using questioner .
  Interpretation Behaviour score(10 questions): good (score>=30 ) moderate (score 21-30) poor (score 0-20).
Nutritional status by body weight | 8 weeks
  To determine changes in BW (body weight in kg) in cancer patients who received cancer-specific ONS compared to those who did not receive ONS after the 8-week intervention. The higher the increase in BW, the better.
Nutritional status by body mass index | 8 weeks
  To determine changes in BMI (body mass index in kg/m2) in cancer patients who received cancer-specific ONS compared to those who did not receive ONS after the 8-week intervention. The higher the increase in BMI, the better.
  BMI is calculated as weight in kilograms divided by the square of the height in meters (kg/m2) and is categorized into four groups according to the cutoff points: underweight (<18.5 kg/m2), normal weight (18.5-22.9 kg/m2), overweight (23-24.9 kg/m2), obese grade 1 (≥25-29 kg/m2) and obese grade 2 (>29 kg/m2)
Nutritional status by haemoglobin | 8 weeks
  To determine changes in Hb (haemoglobin in mg/dL) level in cancer patients who received cancer-specific ONS compared to those who did not receive ONS after the 8-week intervention. The higher the increase in haemoglobin level, the better.
Nutritional status by albumin | 8 weeks
  To determine changes in Albumin level (g/dL) in cancer patients who received cancer-specific ONS compared to those who did not receive ONS after the 8-week intervention. The higher the increase in albumin level, the better

SECONDARY OUTCOMES:
Calorie intake | 8 weeks
  Changes in calorie intake between ONS group vs control group after an 8-week intervention. Assessment of calorie intake using NutriSurvey 2007, Food Recall 2x24h & Food Record 3x24h. The higher subject's calorie (kcal) intake ,the better.
Protein intake | 8 weeks
  Changes in protein intake between ONS group vs control group after an 8-week intervention. Assessment of protein intake using NutriSurvey 2007, Food Recall 2x24h & Food Record 3x24h. The higher subject's protein (gram) intake ,the better
Inflammatory status by CRP | 8 weeks
  The change in inflammatory status between ONS group vs control group assessed by CRP(C-reactive protein in mg/L) level (using CRP Latex Kit) after the 8-week intervention. The lower the value of CRP, the better.
Inflammatory status by IL-1 | 8 weeks
  The change in inflammatory status between ONS group vs control group assessed by IL-1 (interleukin-1 in pg/ml) level (using IL-1 ELISA kit) after the 8-week intervention The lower the value of IL-1, the better.
Inflammatory status by IL-6 | 8 weeks
  The change in inflammatory status between ONS group vs control group assessed by IL-6 (interleukin-6 in pg/ml) level (using IL-6 ELISA kit) after the 8-week intervention. The lower the value of IL-6, the better.
Inflammatory status by TNF-α | 8 weeks
  The change in inflammatory status between ONS group vs control group assessed by TNF-α (Tumor necrosis factor alpha in pg/ml) level (using Kit Quantikine ELISA Human TNF- α) after the 8-week intervention. The lower the value of TNF-α, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Elisna Syahruddin, Phd.MD, Principal Investigator — Persahabatan Hospital
Locations (1):
- Persahabatan General Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Starting December 2023
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal. For more information or to submit a request, please contact: dedyanto.henky@kalbe.co.id